CLINICAL TRIAL: NCT04948541
Title: Effect Of Sleep Apnea Treatment On Temporo-Mandibular Disorders In Patients Suffering From Sleep Apnea
Brief Title: Effect Of Sleep Apnea Treatment On Temporo-Mandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Alessandri Bonetti (Other)
Responsible Party: Sponsor-Investigator, Anna Alessandri Bonetti, Principal Investigator, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3928
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Pain; Pain, Face; Temporomandibular Disorder
Keywords: pain; sleep apnea; temporo-mandibular disorders
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Pain; Facial Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental)
  Interventions: Combination Product: osa treatment
- no treatment (Experimental)
  Interventions: Other: no treatment

INTERVENTIONS:
Combination Product: osa treatment — different treatments can be included
  Arms: treatment
Other: no treatment — no treatment was undergone
  Arms: no treatment

SUMMARY:
Aims of this research are to detect if an improvement in sleep pattern in patients suffering from obstructive sleep apnea (OSA), produces a reduction in pain and dysfunction in the orofacial area by examining variation in temporo-mandibular disorder (TMD) signs and symptoms and if the prevalence of TMDs in OSA patients controlling this disease decreases to levels comparable to healthy subjects.

41 OSA patients will undergo a complete TMD examination prior to start any OSA treatment and after at least 18 months of therapy. Variations in TMD signs and symptoms will be recorded.

DETAILED DESCRIPTION:
Since a bidirectional relationship has been suggested for poor sleep and pain and considering that patients suffering from obstructive sleep apnea (OSA) have been reported to present a higher prevalence of temporo-mandibular disorder (TMD) signs and symptoms compared to healthy controls; aims of this research are to detect if an improvement in sleep pattern in patients suffering from OSA, produces a reduction in pain and dysfunction in the orofacial area by examining variation in TMD signs and symptoms and if the prevalence of TMDs in OSA patients controlling this disease decreases to levels comparable to healthy subjects.

41 OSA patients will undergo a complete TMD examination prior to start any OSA treatment and after at least 18 months of therapy. Variations in TMD signs and symptoms will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from OSA diagnosed by polysomnography not yet undergoing treatment

Exclusion Criteria:

* patients presenting some kind of cognitive impairment, due to difficulties in undergoing TMD examination
* patients presenting dental problems
* patients assuming medications that would alter pain perception
* patients not signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
variation in TMD prevalence according to diagnostic criteria for temporo-mandibular disorders | change from baseline temporo-mandibular disorders at 18 months
  prevalence described as percentage of people having the disease

SECONDARY OUTCOMES:
reduction of TMD signs according to diagnostic criteria for temporo-mandibular disorder | change from baseline temporo-mandibular disorder signs at 18 months
  reduction described as percentage of people resolving the disease
reduction of TMD symptoms according to diagnostic criteria for temporo-mandibular disorder | change from baseline temporo-mandibular disorder symptoms at 18 months
  reduction in pain described by patients through a numeric rating scale going from 0 to 10, were 0 is no pain and 10 is the worst immaginabile pain

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

REFERENCES:
- [Derived] Alessandri-Bonetti A, Lobbezoo F, Mangino G, Aarab G, Gallenzi P. Obstructive sleep apnea treatment improves temporomandibular disorder pain. Sleep Breath. 2024 Mar;28(1):203-209. doi: 10.1007/s11325-023-02883-4. Epub 2023 Jul 25. PMID 37491568